CLINICAL TRIAL: NCT06165380
Title: A Prospective, Multicenter, Phase II Study on the Efficacy and Safety of Cardenilimab Combined With Chemotherapy in the Conversion Therapy of Locally Advanced Esophageal Squamous Cell Carcinoma.
Brief Title: Cardenilimab Combined With Chemotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Li Zhang (Other)
Responsible Party: Sponsor-Investigator, Li Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJCC-EC001
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Squamous Cell Carcinoma; Neoadjuvant Therapies
Keywords: Immunotherapy; Chemotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardenilimab Combined With Chemotherapy (Experimental)
  Interventions: Drug: Cardenilimab Combined With Chemotherapy

INTERVENTIONS:
Drug: Cardenilimab Combined With Chemotherapy — Cardenilimab Combined With Chemotherapy

SUMMARY:
The goal of this trial is to test the efficacy and safety of cardenilimab combined with chemotherapy in the conversion therapy of locally advanced unresectable esophageal squamous cell carcinoma.

type of study: clinical trial

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent before implementing any trial-related procedures; 2. Male or female, age ≥18 years old; 3. Patients with histologically confirmed esophageal squamous cell carcinoma, diagnosed as cT4a, T4b, NXM0 according to the 8th edition of AJCC TNM staging, and assessed as initially unresectable by the surgeon; 4. Have not received any systemic treatment for the current disease in the past, including surgery, anti-tumor radiotherapy, chemotherapy/immunotherapy, etc.; 5. Patients who agree to undergo radical surgical treatment and are judged by the surgeon to have no contraindications to surgery 6. ECOG score 0-1 points; 7. Expected survival time >6 months; 8. With sufficient organ function, subjects must meet the following laboratory indicators:

1. Absolute neutrophil count (ANC) ≥1.5x109/L without using granulocyte colony-stimulating factor in the past 14 days;
2. Without blood transfusion in the past 14 days, platelets ≥100×109/L;
3. Hemoglobin >9g/dL without blood transfusion or erythropoietin use in the past 14 days;
4. Total bilirubin ≤1.5×upper limit of normal (ULN);
5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are within ≤2.5×ULN
6. Serum creatinine ≤1.5×ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥60 ml/min;
7. Good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN;
8. Euthyroid, defined as thyroid stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects can also be enrolled if total T3 (or FT3) and FT4 are within the normal range;
9. Myocardial enzyme spectrum is within the normal range (if the researcher comprehensively judges that simple laboratory abnormalities without clinical significance are also allowed to be included); 9. Female subjects of childbearing potential should receive a urine or serum pregnancy test with a negative result within 3 days before receiving the first dose of study drug (Day 1 of Cycle 1). If a urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Women of non-reproductive age were defined as at least 1 year postmenopausal, or had undergone surgical sterilization or hysterectomy; 10. If there is a risk of pregnancy, all subjects (regardless of male or female) need to use low annual failure rate during the entire treatment period until 120 days after the last dose of study drug (or 180 days after the last dose of chemotherapy drug). Contraceptive measures at 1%.

Exclusion Criteria:

1. Other malignant diseases diagnosed within 5 years before the first dose (excluding radical basal cell carcinoma of the skin, squamous epithelial carcinoma of the skin, and/or carcinoma in situ that has been radically resected);
2. Endoscopically known signs of active bleeding in the lesion;
3. Currently participating in interventional clinical research treatment, or have received other research drugs or used research equipment within 4 weeks before the first dose;
4. Have previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or another type of stimulating or synergistic inhibition of T cell receptors (including but not limited to CTLA-4, OX-40, CD137 etc.) drugs;
5. Have received systemic systemic treatment with Chinese patent medicines with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except for local use to control pleural effusion) within 2 weeks before the first dose;
6. Active autoimmune disease that requires systemic treatment (such as the use of disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred within 2 years before the first dose. Replacement therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatments;
7. Are receiving systemic glucocorticoid treatment (excluding nasal spray, inhaled or other local glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first dose of the study; Note: Physiological doses of glucocorticoids (≤10 mg/day of prednisone or equivalent) are allowed;
8. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
9. People who are known to be allergic to the drugs used in this study;
10. Those with multiple factors that affect capecitabine (such as inability to swallow, intestinal obstruction, etc.);
11. Have not fully recovered from toxicity and/or complications caused by any intervention before initiating treatment (i.e., ≤Grade 1 or reaching baseline, excluding fatigue or alopecia);
12. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
13. Untreated active hepatitis B (defined as HBsAg positivity and a detected HBV-DNA copy number greater than the upper limit of normal value in the laboratory of the research center);

Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

1. The HBV viral load before the first dose is <2500 copies/ml (500 IU/ml), and the subject should receive anti-HBV treatment during the entire study chemotherapy drug treatment period to avoid viral reactivation.
2. Subjects with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-) do not need to receive prophylactic anti-HBV treatment, but need to be closely monitored for viral reactivation 14. Subjects with active HCV infection (HCV antibody positive and HCV-RNA level higher than the lower limit of detection); 15. Get live vaccine within 30 days before the first dose (cycle 1, day 1); NOTE: Injectable inactivated virus vaccine for seasonal influenza is allowed within 30 days before the first dose; however, intranasal live attenuated influenza vaccine is not allowed 16. Pregnant or lactating women; 17. The presence of any serious or uncontrollable systemic disease, such as:

1) The resting electrocardiogram has major abnormalities in rhythm, conduction or morphology that are difficult to control with severe symptoms, such as complete left bundle branch block, second degree or higher heart block, ventricular arrhythmia or atrial fibrillation; 2) Unstable angina, congestive heart failure, New York Heart Association (NYHA) chronic heart failure grade ≥ 2; 3) Any arterial thrombosis, embolism or ischemia occurred within 6 months before selected treatment, such as myocardial infarction, unstable angina, cerebrovascular accident or transient cerebral ischemic attack; 4) Unsatisfactory blood pressure control (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg); 5) There is a history of non-infectious pneumonia requiring glucocorticoid treatment within 1 year before the first dose, or there is currently clinically active interstitial lung disease; 6) Active pulmonary tuberculosis; 7) There is an active or uncontrolled infection that requires systemic treatment; 8) Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction exists; 9) Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis; 10) Poorly controlled diabetes (fasting blood glucose (FBG) >10mmol/L); 11) Those whose urine routine shows urine protein ≥++, and the 24-hour urine protein quantification is confirmed to be >1.0 g; 12) Patients with mental disorders and unable to cooperate with treatment; 18. Evidence of medical history or disease, abnormal treatment or laboratory test values that may interfere with the trial results, prevent the subject from fully participating in the study, or other circumstances that the researcher believes are not suitable for enrollment. The researcher believes that there are other potential risks and are not suitable for participation this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 2-5 years
  The time from randomization to death from any cause.

SECONDARY OUTCOMES:
Pathologic Complete Response | 2-5 years
  According to the detection of pathological specimens after operation, no malignant tumor cells were detected, so the patient achieved complete pathological remission.
Progression-Free-Survival | 2-5 years
  The time between the beginning of treatment and the observation of disease
Overall survival | 2-5 years
  The time from randomization to death from any cause.
Safety | 2-5 years
  The safety of drugs was evaluated from four aspects: adverse events, adverse reactions, serious adverse events and serious adverse reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No